CLINICAL TRIAL: NCT01567878
Title: Ultrasound of Enthesis in Patients With Ankylosing Spondylitis: a Comparative Study With Health Subjects
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Suellen Narimatsu, Principal Investigator, University of Sao Paulo
Other Study IDs: 1649/09
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Spondylitis, Ankylosing
Keywords: ultrasound; MASEI index; clinical and ultrasound correlation; enthesis ultrasound; articular ultrasound; ankylosing spondylitis ultrasound; radiographic and ultrasound correlation
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ankylosing spondylitis: It will be held ultrasound exam in enthesis and joints in patients with ankylosing spondylitis and healthy subjects
- Healthy pelople: It will be held ultrasound exam in enthesis and joints of healthy subjects

SUMMARY:
* Evaluate the correlation of ultrasound MASEI index with clinical, functional, radiographic and laboratorial variables in patients with ankylosing spondylitis.
* Evaluate correlation between articular (shoulders, hips, knees and ankles) ultrasound (synovitis, erosions, power doppler) with same variables.
* Evaluate correlation between articular and enthesis ultrasound exam in this study.
* Compare patients and healthy individuals data, to calculate the ROC curve to estimate predictor value of disease.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis by the Modified New York Criteria (1984)or ASAS classification (2009)
* Healthy people with no history of joint pain, inflammatory lumbar pain inflammatory disease,
* 18 - 65 years old

Exclusion Criteria:

* Fibromyalgia
* Corticosteroid injection in the last 3 months
* Previous surgery in joint or enthesis of study
* Peripheric neuropathy
* Diabetes mellitus
* Hypothyroidism
* Peripheric venous insufficiency (with edema or ocre dermatitis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ankylosing spondylitis healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Ultrasound of enthesis in patients with ankylosing spondylitis: a comparative study with healthy subjects | december
  a comparative study of enthesis by ultrasound revealed statistical differences among patients with ankylosing spondylitis and healthy volunteers in analysis of calcaneal enthesis, plantar fascia and quadriceps.

CONTACTS AND LOCATIONS:
Locations (1):
- Suellen Narimatsu, São Paulo, São Paulo, Brazil